CLINICAL TRIAL: NCT03222934
Title: A Multislice Computed Tomographic Study of the Sphenoid Sinus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Akram Shahat, Dr, Assiut University
Other Study IDs: ASOM
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Nasal Disorder
MeSH Terms: conditions — Nose Diseases | interventions — Multidetector Computed Tomography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nasal disorders: patients with nasal disorders with free sphenoid sinus
  Interventions: Device: multislice computed tomography

INTERVENTIONS:
Device: multislice computed tomography — radiological diagnosis of the status and variations in the sphenoid sinus

SUMMARY:
•Sphenoid sinus is located in the body of sphenoid bone, closed with a thin plate of bone tissue that separates it from the surrounding important structures .Detailed, meticulous preoperative radiological study of sphenoid sinus is the key to successful and safe functional endoscopic sinus surgery and transsphenoidal surgery. The purpose of the study is to delineate the sphenoid sinus radiologically using the multislice computed tomography and to decrease morbidity and mortality during skull base surgeries as the sphenoid sinus is one of the most variable of all sinuses and its relation to vital vascular and nervous elements make its approach a challenge for endoscopic surgeons

DETAILED DESCRIPTION:
Sphenoid sinus is located in the body of sphenoid bone, closed with a thin plate of bone tissue that separates it from the surrounding important structures such as the optic nerve, optic chiasm, cavernous sinus, pituitary gland, and internal carotid artery. Detailed, meticulous preoperative radiological study of sphenoid sinus variations as in Onodi cells (Sphenoethmoidal air cell) is an anatomical variant of the paranasal sinuses, important due to its close proximity to the optic nerve and internal carotid artery. , Pnumatization pattern as the extent of pneumatization is highly variable and potentially jeopardizing to surrounding vital structures , Septation pattern , Intercarotid distance (in millimeters), Bony covering of carotid artery, Bony covering of optic nerve.is the key to successful and safe functional endoscopic sinus surgery and transsphenoidal surgery. The purpose of the study is to delineate the sphenoid sinus radiologically using the multislice computed tomography and to decrease morbidity and mortality during skull base surgeries as the sphenoid sinus is one of the most variable of all sinuses and its relation to vital vascular and nervous elements make its approach a challenge for endoscopic surgeons

ELIGIBILITY:
Inclusion Criteria:

* patients with free sphenoid sinus

Exclusion Criteria:

* pathology in the sphenoid sinus
* refusal of patients for inclusion in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with nasal disorders with free sphenoid sinus
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-04-01 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
The rate of anatomical variations of the sphenoid sinus | 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt